CLINICAL TRIAL: NCT02413099
Title: The Efficacy and Safety of New Herbal Formula (KBMSI-2) in the Treatment of Erectile Dysfunction: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: The Efficacy and Safety of New Herbal Formula (KBMSI-2) in the Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hyun Jun Park (Other)
Responsible Party: Sponsor-Investigator, Hyun Jun Park, Professor, Pusan National University Hospital
Organization: Pusan National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBMSI-2 Study
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — KBMSI-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KBMSI-2 6gm (Experimental): Patients were instructed to take investigational products (KBMSI-2 6g) twice a day for 8weeks at least 1 hour after food intake
  Interventions: Drug: KBMSI-2
- Placebo (Placebo Comparator): Patients were instructed to take placebo twice a day for 8weeks at least 1 hour after food intake
  Interventions: Drug: KBMSI-2

INTERVENTIONS:
Drug: KBMSI-2 — The KBMSI-2 capsules (6gm/capsule) and placebo were provided by Korean Bio Medical Science Institute (Seoul, Korea). KBMSI-2 was analyzed by high-performance liquid chromatography. KBMSI-2 contained major ginsenoside-Rb1: 260.53ug/g, -Rb2: 543.91ug/g, -Rc: 424.92ug/g, -Re: 377.32ug/g, -Rf: 1160.55ug/g, -Rg1: 703.97ug/g, Curcumin 60.73ug/g, Allantoin 98.66ug.g, and Loganin 744.13ug/g. During the study period, two capsules were taken daily for 8 weeks. The placebo capsules were identical in shape, color, and taste.
  Other Names: Better man (brand name)

SUMMARY:
Background: KBMSI-2, which is the herbal formular consisted of Ginseng Radix Rubra, Dioscorea tenuipes, Cornus officinalis Sieb. Et Zucc, Lycium Chinese Mill, Curcuma logna Linn, Honey, improved the erectile function by preserving the smooth muscle content and inhibiting the fibrosis of the corpus cavernosum in STZ-induced diabetic rat model. In this study, the researchers investigated the efficacy and safety of the herbal formula (KBMSI-2) in the treatment of ED.

Material and Methods: Patients were instructed to take investigational products (KBMSI-2 6g or placebo) twice a day for 8 weeks at least 1 hour after food intake. The primary efficacy variable was the change in the EF domain scores of the IIEF questionnaire from baseline. Secondary efficacy measures included change in all domain scores of the IIEF from baseline, change in question 2 and 3 of the SEP2,3, from baseline.

ELIGIBILITY:
Inclusion criteria were as follows:

* men with history of ED for at least 6 months according to the National Institutes of Health (NIH) Consensus Statement (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance);
* erectile function (EF) domain scores of the International Index of Erectile Function (IIEF) questionnaire ≤ 25;
* age range between 19 and 40 years old;
* patients were required to be involved in a stable, monogamous relationship with a female sexual partner and having failed >50% of at least four sexual attempts during the run-in period.

Exclusion criteria were as follows:

* Men with the following conditions were excluded from the study:
* penile anatomical defects,
* spinal cord injury,
* radical prostatectomy,
* and radical pelvic surgery;
* a primary diagnosis of another sexual disorder;
* uncontrolled DM (HBA1C> 12%);
* serum creatinine>2.5mg/dL;
* major uncontrolled psychiatric disorder;
* history of major hematological, renal, or hepatic abnormalities;
* recent (within the previous 6 months) history of cardiovascular disease, stroke or myocardial infarction, cardiac failure, unstable angina, life-threatening arrhythmia and a history of alcoholism or substance abuse.
* Patients having taken PDE5 inhibitors and testosterone replacement therapy within 2 weeks were excluded in the study. Concomitant use of ED treatment was forbidden.

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2013-01-03 (Actual)

PRIMARY OUTCOMES:
Change in the EF domain scores of the IIEF questionnaire from baseline | Baseline, 4weeks, 8weeks
  calculated by comparing total scores from questions 1 to 5 and 15 from IIEF questionnaire

SECONDARY OUTCOMES:
Change in all domain scores of the IIEF from baseline | Baseline, 4weeks, 8weeks
change in question 2 and 3 of the Sexual Encounter Profile (SEP2: Were you able to insert your penis in your partner's vagina? SEP3: Did your erection last long enough for you to have a successful intercourse?) from baseline | Baseline, 4weeks, 8weeks
  change in question 2 and 3 of the Sexual Encounter Profile (SEP2: Were you able to insert your penis in your partner's vagina? SEP3: Did your erection last long enough for you to have a successful intercourse?) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Pusan National University Hospital, Busan, South Korea